CLINICAL TRIAL: NCT03192800
Title: Clinical Outcome in Patients With Spinal Dural Arteriovenous Fistulas
Brief Title: Clinical Outcome in Patients With Spinal Dural Arteriovenous Fistulas (COPSDAVF)
Acronym: COPSDAVF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hongqi Zhang, MD (Other)
Collaborators: Beijing Haidian Hospital (Other)
Responsible Party: Sponsor-Investigator, Hongqi Zhang, MD, Director, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Other Study IDs: COPSDAVF
Record Dates: First submitted 2017-06-14; First posted 2017-06-20 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Spinal Vascular Disorder Nos
Keywords: clinical outcome; prognositic factor; spinal dural arteriovenous fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Spinal dural arteriovenous fistulas (SDAVFs) are the most common vascular disorder of the spine and account for approximately 70% of spinal vascular malformation.They are a rare pathology with an excepted incidence of only 5-10 new cases per million inhabitants per year. Most fistulas are found in the thoracolumbar region and > 80% of all SDAVFs are located between T6 and L2, whereas the cranio-cervical, cervical and sacral fistulas are more rare. SDAVFs have an overwhelmingly male predominance (80%), with an age presentation in the fifth or sixth dacede. It is presumed that SDAVFs are acquired diseases. A typical SDAVF is located inside the dural mater close to nerve root. It is fed by a radiculomeningeal artery and enters a radicular vein that merges in the perimedullary plexus. The presence of a shunt leads to a reversal of blood flow to the spinal cord venous system, which then induces venous hypertensive myelopathy.

DETAILED DESCRIPTION:
The initial symptoms of venous congestion include gait disturbances, sensory symptoms (hyperesthesia and paresthesia), and sphincter dysfunction. These neurological symptoms are unspecific, so SDAVFs often go clinically underdiagnosed or misdiagnosed. But SDAVFs typically demonstrated a characteristic imaging appearance on spinal MRI including multilevel centromedullary cord T2 hyperintensity, enlarged intradural vessels along the dorsal and ventral aspect of the cord. If an SDAVF is suspected, conventional spinal angiography is required to confirm the diagnosis and determine the location of the fistula. Flowing diagnosis, expedient treatment is required, both microsurgery and endovascular embolization are safe and can achieve complete occlusion, the progression of the neurological deficits can be stopped in most instances.

However, it is difficult to predict whose symptoms will improve and whose will stabilize or deteriorate. Due to the low incidence of the SDAVFs, nearly all studies which have been published about the clinical outcome and prognostic factors of SDAVFs are relatively limited and most of them are retrospective. In these studies, the preoperative severity of disability, age, gender, location of fistula and duration of symptoms have been analyzed as prognostic factors, therefore it remains unclear which are the most reliable predictor of clinical outcome. Moreover, the conclusions may be biased by long span of follow-up period or few clinical cases. Besides, the fitulas at the craniocervical junction often present with hemorrhage, while those below conus constitute 3 types of lesions. So the invsetigator conduct this prospective cohort study to clarify the 1-year outcome of patients with cervical and thoracolumbar SDAVFs and to determine the main prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* patient diagnosed with spinal dural arteriovenous fiatulas
* the fiatula locate between C2 and L5
* patient not received surgical or interventional treatment before
* patient with normal cardiac, renal and hepatic function
* patient capable of understanding the content of the patient information / Informed Consent Form
* patient willing and able to participate in the registry

Exclusion Criteria:

* patient received surgical treatment or interventional treatment before
* patient is pregnant patient allergic to iodine
* patient unable to complete follow-up
* patient with cerebral lesions patient with other spinal lesions
* patient with cardiac, renal or hepatic dysfunction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with spinal dural arteriovenous fistulas admitted to department of neurosurgery in Xuanwu Hospital and department of neurosurgery in Beijing Haidian Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-03-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of the spinal cord function | 1 day before operation and 3 months, 6 months, 12 months postoperation
  Modified Aminoff & Logue's Scale for evaluating the spinal cord function

SECONDARY OUTCOMES:
Modified Denis Pain and Numbness Scale (mDPNS) | 1 day before operation and 3 months, 6 months, 12 months postoperation
  mDPNS for evaluating the sensory function of patients with SDAVFs before and after operations

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Hongqi, MD.PHD., Study Director — Xuanwu Hospital, Beijing
Locations (1):
- Neurosurgery Department of Xuanwu hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cenzato M, Versari P, Righi C, Simionato F, Casali C, Giovanelli M. Spinal dural arteriovenous fistulae: analysis of outcome in relation to pretreatment indicators. Neurosurgery. 2004 Oct;55(4):815-22; discussion 822-3. doi: 10.1227/01.neu.0000137630.50959.a7. PMID 15458589
- [Result] Steinmetz MP, Chow MM, Krishnaney AA, Andrews-Hinders D, Benzel EC, Masaryk TJ, Mayberg MR, Rasmussen PA. Outcome after the treatment of spinal dural arteriovenous fistulae: a contemporary single-institution series and meta-analysis. Neurosurgery. 2004 Jul;55(1):77-87; discussion 87-8. doi: 10.1227/01.neu.0000126878.95006.0f. PMID 15214976
- [Result] Fugate JE, Lanzino G, Rabinstein AA. Clinical presentation and prognostic factors of spinal dural arteriovenous fistulas: an overview. Neurosurg Focus. 2012 May;32(5):E17. doi: 10.3171/2012.1.FOCUS11376. PMID 22537126
- [Result] Sherif C, Gruber A, Bavinzski G, Standhardt H, Widhalm G, Gibson D, Richling B, Knosp E. Long-term outcome of a multidisciplinary concept of spinal dural arteriovenous fistulae treatment. Neuroradiology. 2008 Jan;50(1):67-74. doi: 10.1007/s00234-007-0303-4. Epub 2007 Nov 20. PMID 18026943
- [Result] Saladino A, Atkinson JL, Rabinstein AA, Piepgras DG, Marsh WR, Krauss WE, Kaufmann TJ, Lanzino G. Surgical treatment of spinal dural arteriovenous fistulae: a consecutive series of 154 patients. Neurosurgery. 2010 Nov;67(5):1350-7; discussion 1357-8. doi: 10.1227/NEU.0b013e3181ef2821. PMID 20871454
- [Result] Krings T, Geibprasert S. Spinal dural arteriovenous fistulas. AJNR Am J Neuroradiol. 2009 Apr;30(4):639-48. doi: 10.3174/ajnr.A1485. Epub 2009 Feb 12. PMID 19213818